CLINICAL TRIAL: NCT05623254
Title: Feasibility and Effectiveness of a Mindfulness Program Delivered by Web to Patients During Hospitalization and Caregivers: a Pilot Study (KMPO Project)
Brief Title: Feasibility and Effectiveness of a Mindfulness Program Delivered by Web to Patients During Hospitalization and Caregivers.
Acronym: KIMPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KIMPO
Record Dates: First submitted 2022-10-28; First posted 2022-11-21 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Chronic Migraine; Multiple Sclerosis; Motoneuron Disease
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: A pilot, prospective, interventional, monocenter study
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAU + MINDF (Treatment-as -Usual + Mindfulness) (Other): Treatment-as-usual combined with weekly mindfulness sessions delivered on-line for patients and caregivers (a specific platform for on-line sessions will be used)
  Interventions: Other: no comparator - TAU (Treatment-as-usual)

INTERVENTIONS:
Other: no comparator - TAU (Treatment-as-usual) — Learning the ability in mindfulness practice by specific measure (FFMQ) changes in FIVE FACET MINDFULNESS QUESTIONNAIRE (FFMQ) compared to baseline): this questionnaire measures the mindfulness ability of patients before and after the APP application (minimum score 113.7-low mindfulness ability=worse outcome ; maximum score 144.3-high mindfulness ability=better outcome) [Time Frame: At Three-six months]
  Introduction of the mindfulness program during a preliminary face-to-face session to patients and caregivers
  TAU Weekly mindfulness sessions delivered on-line for patients and caregivers (a specific platform for on-line sessions will be used)

SUMMARY:
Hospitalization is often a traumatic event so stressful for the life of patients. Isolation, loneliness, worries about clinical examinations, results from examinations and final diagnosis, uncertainty about the future are the most common feelings that patients report when during hospitalized for different disease conditions; these feelings are not related to the pathological condition.

Also the discomfort of the caregivers is significant, as the necessities and priorities of the family change significantly during the hospitalization of a member (worries about the future, help and support are not enough to sustain the situation, problems with the work schedule ). Nowadays in North American and North European countries, mindfulness practice is offered to patients by multifaith Chaplaincy teams and health-care operators (e.g. physicians, nurses, psychologists), as a way of helping patients come to terms with diagnosis and adjust to their prognosis. To the extent that patients can bear it, instructions are given to keep coming back to the present moment, here and now, to bodily and affective experience, relaxing in it. To that purpose patients are encouraged to accept the situation as it develops, and let go of excessive concerns and unhelpful narratives that undermine the capacity to manage pain, fear and suffering. Moreover, similar programmes are designed for caregivers and the patients' families, aimed at developing their resilience in delivering the support, via face-to-face sessions, and instructions and encouragement for a regular practice at home.

In the last years, due to the dramatic emergency for the COVID-19 pandemic, different applications for mindfulness have been realized by specific APPs or web platforms that allow patients to practice mindfulness regularly guided by a physician or an expert in mindfulness: patients can stay at home and mindfulness sessions can be delivered by technological modalities. In different hospitals, protocols have been implemented for the treatment of patients remotely, using specific platforms or APPs. These remote interventions are complementary to the regular face-to-face sessions and they are suitable for most patients and easily applied.

DETAILED DESCRIPTION:
Background: Hospitalization is often a traumatic event so stressful for the life of patients. Isolation, loneliness, worries about clinical examinations, results from examinations and final diagnosis, uncertainty about the future are the most common feelings that patients report when they are hospitalized for different disease conditions; these states of mind may be experienced independently of the type of pathological condition they are affected by Also the discomfort of the caregivers is significant, as the necessities and priorities of the family change significantly during the hospitalization of a member (worries about the future, help and support are not enough to sustain the situation, problems with the work schedule ) Significance: The practice of mindfulness has become common in different clinical applications, pain, anxiety and other kinds of disease. In particular protocols based on mindfulness practice are often combined to pharmacological therapies, as initial findings support the utility of mindfulness intervention to modulate attention and emotional reactions to pain chronification Meditation has a long history of use for increasing calmness and physical relaxation, improving psychological balance, coping with illness, and enhancing overall health and well-being. The practice has the purpose to teach individuals how to maintain focus on a stimulus while simultaneously allowing intruding thoughts/feelings to be acknowledged, but not judged.

Hospitalization is often a traumatic event so stressful for the life of patients. Isolation, loneliness, worries about clinical examinations, results of examinations and final diagnosis, uncertainty about the future are the most common feelings that patients report during hospitalization for different disease conditions; these states of mind may be experienced independently of the type of pathological condition the patients are affected by.

Also the discomfort of the caregivers is significant, as the necessities and priorities of the family change significantly during the hospitalization of a member (worries about the future, help and support are not enough to sustain the situation Nowadays in North American and North European countries, mindfulness practice is offered to patients by multifaith Chaplaincy teams and health-care operators (e.g. physicians, nurses, psychologists), as a way of helping them come to terms with the diagnosis and adjust to their prognosis. To the extent that they can bear it, instructions are given to keep coming back to the present moment, here and now, to bodily and affective experience, relaxing in it. To that purpose patients are encouraged to accept the situation as it develops, and let go of excessive concerns and unhelpful narratives that undermine the capacity to manage pain, fear and suffering.

Moreover, similar programmes are designed for caregivers and the patients' families, aimed at developing resilience in delivering their support, via face-to-face sessions, and instructions and encouragement for a regular practice at home.

In the last years, due to the dramatic emergency for the COVID-19 pandemic, different applications for mindfulness have been realized by specific APPs or web platforms that allow patients to practice mindfulness regularly guided by a physician or an expert in mindfulness: patients can stay at home and mindfulness sessions can be delivered by technological modalities.

In several hospitals, different protocols have been implemented for the treatment of patients remotely, using specific platforms or APPs. These remote interventions are complementary to the regular face-to-face sessions and they are suitable for most patients and easily applied.

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 18 and 70 yrs; patients hospitalized at our neurological department; patients at the day hospital service

Patients (age from 18 to 70 yrs) hospitalized suffering from: Chronic migraine with medication overuse; Neuropathic Pain; Multiple Sclerosis are included into the project and caregivers

Exclusion Criteria:

patients not able to understand the italian language; patients with confirmed psychiatric comorbidities; patients who are not able to understand the consent module form and sign it; (or patients with mental capacity issues)

Caregivers aged between 18-70 yrs old, will be admitted into the study if they fall in the 18-70 years age bracket, and understand the Italian language , in the absence of psychiatric conditions (reported specific therapy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
MINDFULNESS | Three-six months
  Learning the ability in mindfulness practice by specific measure (FFMQ) changes in FIVE FACET MINDFULNESS QUESTIONNAIRE (FFMQ) compared to baseline): this questionnaire measures the mindfulness ability of patients before and after the APP application (minimum score 113.7-low mindfulness ability=worse outcome ; maximum score 144.3-high mindfulness ability=better outcome) [Time Frame: At Three-six months]

CONTACTS AND LOCATIONS:
Overall Officials: Licia MI Grazzi, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroalgology Unit, Milan, Italy

IPD SHARING:
Plan to Share IPD: No